CLINICAL TRIAL: NCT00006199
Title: Study of the Farnesyl Transferase Inhibitor, R115777, in Combination With Topotecan (NYU 99-32)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Purpose: Treatment
Other Study IDs: NCRR-M01RR00096-1001; M01RR000096 (NIH)
Record Dates: First submitted 2000-09-09; First posted 2000-09-11 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-01

CONDITIONS: Cancer
Keywords: solid tumor
MeSH Terms: conditions — Neoplasms | interventions — tipifarnib; Topotecan

INTERVENTIONS:
Drug: R115777 (farnesyl transferase inhibitor)
Drug: Topotecan

SUMMARY:
The purpose of this clinical trial is to establish the safest doses for the combination of a farnesyl transferase inhibitor, R115777 plus topotecan in patients with advanced solid tumors, previously treated or beyond standard therapy of clinical benefit. Maximum tolerated dose, dose limiting toxicity and the activity of this combination will be assessed.

This chemotherapy regimen is a two-pronged attack at the way cancer cells replicate. R115777 is a compound that may inhibit cancer cell growth by interfering with the p21 ras oncogene, while topotecan, a topoisomerase-1 inhibitor, works on cancer cells not subject to control by the ras oncogene. Animal studies suggest that the combination may be synergistic. Another advantage is that R115777 can be taken by mouth.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced solid tumors with previous treatment or beyond standard therapy of significant clinical benefit
* Therapy with no more than 3 prior chemotherapy regimens
* Radiotherapy to less than 25% of bone marrow volume (no pelvic radiation)
* Adequate organ function
* Recovery from the effects of prior chemotherapy and radiation therapy, with at least a 4 week interval. All prior toxicities should have resolved to baseline prior to entry into the study.
* Good performance status
* Anticipate life expectancy of at least 6 months
* Not pregnant or lactating.
* Sexually active men and women of childbearing age must use adequate contraception.
* Be able to give signed, written informed consent.
* No gastrointestinal condition that could affect the absorption of the drug
* No active infection requiring systemic medical therapy one week prior to chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- NYU Cancer Institute, New York, New York, United States